CLINICAL TRIAL: NCT03915431
Title: A Phase 1/2 Randomized Study to Evaluate the Safety and Tolerability of Intracarotid Artery Administration of NCS-01 in Patients With Acute Ischemic Stroke
Brief Title: A Study of NCS-01 in Patients With Acute Ischemic Stroke
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NC Medial Research Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCS-01-01
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NCS-01 (Experimental): human bone marrow derived cells
  Interventions: Biological: NCS-01
- sham (Sham Comparator): sham procedure
  Interventions: Biological: NCS-01

INTERVENTIONS:
Biological: NCS-01 — single infusion

SUMMARY:
This is an initial Phase1/2 dose-finding, randomized, multi-center study to evaluate the safety and tolerability of NCS-01 in patients with acute ischemic stroke. All patients will be randomized within 48 hours of stroke onset. This study will be conducted in 2 stages.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18 to 85 years inclusive
* Clinical evidence of acute ischemic unilateral cerebral infarction
* - Evidence of neurologic deficits as defined by NIHSS 6 to 18 or NIHSS < 6 with Fugl-Meyer upper extremity subtotal 6 to 40 inclusive
* Women of child bearing potential who agrees to take acceptable birth control as described in the ICF
* Provide written informed consent before participation, either by patient or a legal representative

Exclusion Criteria:

* Progressive neurologic deficit
* An inability to undergo an MRI scan
* Any malignancies within the last 5 years
* Previous organ transplantation
* Participation in another clinical trial with an investigational drug, device or biologic within the preceding 3 months
* Women of childbearing potential with a positive pregnancy test
* Already dependent in activities of daily living (Rankin scale 3 or more) before the present acute stroke
* Known hypersensitivity, allergy or intolerance to the similar biologic interventions
* Any other clinically relevant acute or chronic diseases which could interfere with patients' safety during the trial, or expose them to undue risk, or which could interfere with study objectives judged by Investigator based on medical history, physical examination, laboratory tests and/or ECG

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events -Safety by Incidence of Treatment-Emergent Adverse Events | multiple times for the duration of the study (baseline through Month 12)
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0" . Incidence and nature of adverse events; vital signs;
National Institutes of Health Stroke Scale (NIHSS) | 1 hour, 3 hours, and 6 hours post infusion
  Change from baseline in the NIHSS NIHSS is a systematic assessment tool that provides a quantitative measure of stroke-related neurologic deficit. The score for each ability is a number between 0 and 4, 0 being normal functioning and 4 being completely impaired. The patient's NIHSS score is calculated by adding the number for each element of the scale; 42 is the highest score possible. In the NIHSS, the higher the score, the more impaired a stroke patient is.
Number of participants with change in in physical examination | multiple times from baseline through Month 12
  physical examination changes General appearance ,Head, eyes, ears, nose, and throat, Respiratory, Cardiovascular, Musculoskeletal, Abdomen, Neurologic, Extremities, Dermatologic, Lymphatic)
Number of participants with change in Electrocardiography (ECG) | multiple times for the duration of the study (baseline through Month 12)
  ECG (standard digital 12-lead in singlicate)
Number of participants with change in clinical laboratory evaluations | multiple times for the duration of the study (baseline through Month 12)
  changes in clinical laboratory evaluations (Creatinine, Potassium(K+),Sodium (Na+) , Chloride (Cl-), Magnesium (Mg++), Calcium, Inorganic phosphate, Glucose, Urea,Bilirubin (Total) ,Bilirubin (direct), AST, ALT, GGT, Alkaline phosphatase, Total Protein Albumin,

SECONDARY OUTCOMES:
Number of participants with change in Modified Rankin Scale (mRS) | multiple times for the duration of the study (baseline through Month 12)
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke.Score Description 0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Number of participants with change in Cytokine panel (IL-1, 6, 8, etc.) | multiple times for the duration of the study (baseline through Month 12)
  blood test for proteins that modulate the inflammatory response
Number of participants with change in MRI | multiple times for the duration of the study (baseline through Month 12)
  global white matter and grey matter volumetrics; cortical thinning on MRI
Number of participants with change in Barthel Index | multiple times for the duration of the study (baseline through Month 12)
  Barthel Index is a 4 point scale of Activities of Daily Living

OTHER OUTCOMES:
Number of participants with change in Domain-specific Scales (Fugl-Meyer) | multiple times for the duration of the study (baseline through Month 12)
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, sensation, balance, joint range of motion and joint pain in patients with post-stroke hemiplegia (Fugl-Meyer, Jaasko, Leyman, Olsson, & Steglind, 1975; Gladstone, Danells, & Black, 2002). It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Savitz, md, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No